CLINICAL TRIAL: NCT04732676
Title: Efficacy of a Smartphone App Designed to Manage Craving and Individual Predictors of Substance Use / Addictive Behavior Among Individuals With Addictive Disorders
Brief Title: Efficacy of a Smartphone App. Designed to Manage Craving & Individual Predictors of Substance Use/Addictive Behavior
Acronym: CRAVINGMANAGER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2020-A01707-32
Record Dates: First submitted 2019-05-10; First posted 2021-02-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Addiction
Keywords: craving
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial comparing two parallel groups. This is a comparative study of superiority that evaluates the efficacy of using an interventional smartphone application,in reducing main problematic substance use/addictive behavior after 4 weeks, and after 4 months among participants requesting treatment for substance or behavioral addiction.
Who Masked: Participant, Care Provider, Investigator
Masking Description: After randomization, the application will be installed on participant's smartphone (or smartphone loaned for the study).
  Randomization code will unlock one of the 2 versions of the application:
  * Restricted version (only EMA) for control group
  * Full interventional (active) version (EMA + EMI) for experimental group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): participants will receive and use during 4 weeks the full interventional version of the smartphone application (combining EMA + EMI) targeting craving and personal situations at risk for use
  Interventions: Other: Smartphone application
- control group (Placebo Comparator): : participants will receive and use a restricted version of the smartphone application (only EMA: 4 electronic questionnaires per day to assess main problematic substance use / addictive behavior) during 4 weeks
  Interventions: Other: Smartphone application

INTERVENTIONS:
Other: Smartphone application — Ecological Momentary Assessment (EMA)
  : ambulatory assessment of behaviors/symptoms in real-time on smartphones

SUMMARY:
Test the Efficacy of a smartphone application designed to manage craving and individual predictors of substance use / addictive behavior among individuals with addictive disorders

DETAILED DESCRIPTION:
This translational project is the clinical application of research results from the University of Bordeaux, Sanpsy Lab, CNRS USR3413 - on individual predictors of substance use. This project will test the efficacy of a smartphone application to help subjects concerned about reducing or stopping their substance use / behavioral addiction.

This new therapeutic tool, designed by University of Bordeaux, Sanpsy Lab, CNRS USR3413 - to manage craving and individual predictors of use, will offer the possibility of an easy to-use and personalized intervention accessible to the greatest number of subjects.

Based on our previous results that supports that, for all types of addiction, craving and individual cues are a significant drive for use in people with addiction, the application tested in this study was designed to be used among people presenting various types of addiction (substance and behavioral addictions). The application will also evaluate all concurrent substance uses and addictive behaviors to identify and prevent risk of addiction transfers.

ELIGIBILITY:
Inclusion Criteria:

* Participants requesting help for substance or behavioral addiction in one of the participating specialized addiction treatment centers, and with more than 1-month-delay before treatment admission
* Age >= 18 years of age
* With at least one substance or behavioral addiction (DSM-5 criteria)
* Affiliated person or beneficiary of a social security scheme.
* Free, informed and written consent signed by the participant and the investigator

Exclusion Criteria:

* Medical, psychiatric or addiction condition that warrants immediate treatment intervention
* Patients with somatic, cognitive or other disorders preventing the use of the device (deafness, impaired vision, illiteracy....)
* Difficulty in understanding and / or writing French
* Not familiar with the use of smartphone
* Individuals participating in another study that includes an ongoing exclusion period
* Be deprived of liberty due to an ongoing legal procedure
* Individuals under legal protection
* Be under guardianship or under curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
The decrease of main problematic substance use / addictive behavior | 4 weeks
  We will compare the percentage of participants for whom a 20% decrease in main problematic substance use / addictive behavior was observed between 1st week and 4 th week of smartphone application use in the experimental group versus the control group

SECONDARY OUTCOMES:
Efficacy of the intervention in reduction on addiction severity (ASI) and craving for primary addiction, | At 1-month and 4-month follow-up
  Multifactorial addiction severity ASI "Composite Score" for the main problematic addiction (drug or alcohol or tobacco or behavioral addiction) : Range 0-1 (1: higher severity) and craving self-reported in the last EMA week, and reported in the Craving evaluation scale developed by the University of Bordeaux Addiction Team of the Sanpsy Laboratory will be used. It is an heteroevaluation of craving for all substances and addictive behaviors reported by the subject. This tool explores the frequency of craving, corresponding to the number of days craving was reported during the last 30 days, as well as mean and maximum intensity on a scale ranging from 0 (no craving) to 10 (extreme craving).
  Comparison between baseline, 1-month et 4-month follow-ups of frequency, mean and maximum intensity of craving for main problematic addiction
Factors associated with application efficacy among initial addiction severity (ASI), initial craving for primary addiction, type of primary addiction, comorbid psychiatric disorders (MINI), and addiction treatment (ASI and TSR) | inclusion
  Evaluation of the initial severity of addiction ASI "Composite Score" for the main problematic addiction (drug or alcohol or tobacco or behavioral addiction) : Range 0-1 (1: higher severity), initial craving frequency and intensity with craving evaluation scale, the type of addiction,comorbid psychiatric disorders (evaluated with Mini International Neuropsychiatric Interview), and past or concomitant addiction treatment (evaluated by ASI and Treatment Service Review).
Temporal evolution of craving and substance use/addictive behaviors The evolution and temporal trajectories of craving intensity, substances use/addictive behaviors measured with EMA in daily life | 4 weeks
  During the 4 weeks use of the application, all participants will be instructed to complete 4 daily EMA electronic interviews to assess craving-and substance use/addictive behavior (see Serre, Fatseas et al. 2012). At each electronic interview, participants will be asked to rate the maximum level of craving (i.e. the desire to use the main substance/addictive behavior) that they felt since the previous assessment on a seven-point scale (1 no desire to 7 extreme desire), and will also be asked if they had used, since the previous assessment, the main substance/addictive(yes/no)
  - The evolution and temporal trajectories of substances use/addictive behaviors measured with EMA in daily life
Feasibility of the smartphone application as assessed by use of the app (EMA responses) and drop-out rates | at 1-month
  Feasibility will be assessed at the 1-month follow-up by number of days and frequency of use of the application (calculated from EMA responses: number of questionnaires answered on total number of questionnaires proposed by the application), rate of participants not completing the study, and reasons for stopping
Acceptability of the smartphone app assessed by AES, D-WAI and u-MARS | at 1-month
  Acceptability will be assessed at 1-month follow-up with AES, D-WAI and uMARS. The Acceptability E-scale (AES) is a 6-item questionnaire that evaluates the extent to which subjects find E-health systems acceptable. Each item is ranked on a 5-point Likert scale, generating a total score of acceptability ranging from 6 (lowest acceptability) to 30 (highest acceptability) (Micoulaud-Franchi, Sauteraud et al. 2016). The Digital Working Alliance Inventory (D-WAI) measures factors (goals, tasks and bond) to examine the therapeutic relationship between the participant and the app (Henson et al., 2019). The user version of the Mobile Application Rating Scale (uMARS) is a simple tool that can be reliably used by end-users to assess the quality of mHealth apps (Stoyanov et al., 2016).
Impact on subsequent standard treatment at 4-month follow -up | at 4-month follow-up
  Impact of the 4 weeks use of the smartphone application Potential impact (positive or negative) of the 4 weeks use of the smartphone application on subsequent treatment will be assessed at 4-month follow-up with rate of first-time attendance to the standard treatment, time to first-time attendance to the standard treatment, compliance with standard treatment (Treatment Service Review), and evolution of severity of addiction during the standard treatment (ASI Composite Score). Follow-ups measures will be compared to baseline measures, and the difference will be compared between the two groups.
Acceptability of the smartphone app assessed by AES, D-WAI and u-MARS | at 1-mont
  Intervention Satisfaction will be assessed at 1-month follow-up with the Client Satisfaction Questionnaire (CSQ-8), that is a multi-item measure of satisfaction related to healthcare (Larsen et al., 1979; Kapp et al., 2014). The CSQ-8 total score ranges from 8 to 32. A higher score represents greater satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: MARC AURIACOMBE, MD, Prof, Principal Investigator — Centre Hospitalier CHARLES PERRENS
Locations (1):
- Centre Hospitalier Charles PERRENS, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serre F, Moriceau S, Donnadieu L, Forcier C, Garnier H, Alexandre JM, Dupuy L, Philip P, Levavasseur Y, De Sevin E, Auriacombe M; for Craving-Manager RCT investigator group. The Craving-Manager smartphone app designed to diagnose substance use/addictive disorders, and manage craving and individual predictors of relapse: a study protocol for a multicenter randomized controlled trial. Front Psychiatry. 2023 May 15;14:1143167. doi: 10.3389/fpsyt.2023.1143167. eCollection 2023. PMID 37255691